CLINICAL TRIAL: NCT02826850
Title: Comparative Study of Neurotomy by Radiofrequency of Genicular Nerves, Guided by Fluoroscopy, and Neurotomy by Radiofrequency of Saphenous Nerve, Guided by Ultrasound, for the Treatment of Chronic Knee Pain in Patients With Osteoarthritis .
Brief Title: Saphenous Nerve Radiofrequency for Knee Osteoarthritis Trial
Acronym: SAPHENERO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, M.D., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 55153516.0.0000.0068
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Pulsed Radiofrequency Treatment; Ultrasonography, Interventional
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genicular nerves (Sham Comparator): Neurotomy by radiofrequency of genicular nerves knee guided by fluoroscopy
  Interventions: Procedure: Genicular nerves
- Saphenous Nerve (Active Comparator): Neurotomy of saphenous nerve by radiofrequency on the distal third of the thigh, guided by ultrasound
  Interventions: Procedure: Saphenous Nerve

INTERVENTIONS:
Procedure: Saphenous Nerve — Saphenous nerve neurotomy by radiofrequency, guided by ultrasound.
  Arms: Saphenous Nerve
Procedure: Genicular nerves — Genicular nerves neurotomy by radiofrequency, guided by fluoroscopy
  Arms: Genicular nerves

SUMMARY:
This project is one of four components of a thematic project that aims to evaluate the use of ultrasound in regional and infiltration blocks, called "Use of ultrasound in regional blocks and infiltration for the treatment of acute and chronic pain".

It aims to evaluate quantitatively and qualitatively the knee pain control in patients with osteoarthritis after neurotomy by saphenous nerve radiofrequency guided by ultrasound , compared to neurotomy by radiofrequency of genicular nerves guided by fluoroscopy .

Differences between total consumption of analgesics, side effects of medications , impact on quality of life and functional capacity in patients undergoing saphenous nerve neurotomy by radiofrequency guided by ultrasound compared to neurotomy by radiofrequency of genicular nerves guided by fluoroscopy, will also be evaluated.

DETAILED DESCRIPTION:
BACKGROUND: Osteoarthritis of the knees is currently a major public health problem, with patients suffering from pain and functional limitation. Depending on the severity of the impairment, the definitive treatment is surgical, but the old ages often associated and morbidities present in these patients some times limit such conduct. More effective treatments for pain control are necessary.

OBJECTIVES: To evaluate quantitative and qualitative pain control in patients with osteoarthritis in knees after neurotomy of saphenous nerve by radiofrequency guided by ultrasound, compared to neurotomy by radiofrequency of genicular nerves guided by fluoroscopy.

METHODS: This was a prospective, randomized clinical study and blind to the evaluators. Will include 20 patients with knee osteoarthritis grade III or IV, refractory to medical treatment. A group will be submitted to neurotomy by radiofrequency of genicular nerves guided by fluoroscopy and the other group will receive neurotomy by radiofrequency of saphenous nerve, guided by ultrasound. They will be assessed in pain intensity at rest and movement, functionality, satisfaction and adverse effects related to treatment. Patients will be evaluated 15 days, 1 month, 3, 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Will be included patients older than 18 years, who have moderate to strong chronic pain in knee on most of the days days for at least 3 months, with osteoarthritis of the knee documented by graded radiologically at 3 to 4 in Kellgren-Lawrence rating, refractory to medical treatment (physical therapy, oral analgesics, intra-articular injections of hyaluronic acid or corticosteroids).

Exclusion Criteria:

* The exclusion criteria are: acute knee pain, prior surgery on the knee, another connective tissue disease affecting the knee, psychiatric or neurological disorders, intra-articular injection of hyaluronic acid or corticosteroid for less than 3 months, pain related to nerve sciatic, use of anticoagulants and pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 90 days
  Number verbal scale

SECONDARY OUTCOMES:
Opioids consumption | 90 days
  Morphine oral equivalent dose needed
Side effects | 90 days
  Nausea, vomiting, sedation
Functional capacity | 90 days
  WOMAC score

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Ashmawi, Ph.D, Principal Investigator — Head of the Pain Management Unit; Joaquim E Vieira, Ph.D, Principal Investigator — Associated Professor of Anesthesiology Department
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Andrianakos AA, Kontelis LK, Karamitsos DG, Aslanidis SI, Georgountzos AI, Kaziolas GO, Pantelidou KV, Vafiadou EV, Dantis PC; ESORDIG Study Group. Prevalence of symptomatic knee, hand, and hip osteoarthritis in Greece. The ESORDIG study. J Rheumatol. 2006 Dec;33(12):2507-13. PMID 17143985
- [Background] Mannoni A, Briganti MP, Di Bari M, Ferrucci L, Costanzo S, Serni U, Masotti G, Marchionni N. Epidemiological profile of symptomatic osteoarthritis in older adults: a population based study in Dicomano, Italy. Ann Rheum Dis. 2003 Jun;62(6):576-8. doi: 10.1136/ard.62.6.576. PMID 12759299
- [Background] Felson DT, Naimark A, Anderson J, Kazis L, Castelli W, Meenan RF. The prevalence of knee osteoarthritis in the elderly. The Framingham Osteoarthritis Study. Arthritis Rheum. 1987 Aug;30(8):914-8. doi: 10.1002/art.1780300811. PMID 3632732
- [Background] Ikeuchi M, Ushida T, Izumi M, Tani T. Percutaneous radiofrequency treatment for refractory anteromedial pain of osteoarthritic knees. Pain Med. 2011 Apr;12(4):546-51. doi: 10.1111/j.1526-4637.2011.01086.x. Epub 2011 Apr 4. PMID 21463469
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Akbas M, Luleci N, Dere K, Luleci E, Ozdemir U, Toman H. Efficacy of pulsed radiofrequency treatment on the saphenous nerve in patients with chronic knee pain. J Back Musculoskelet Rehabil. 2011;24(2):77-82. doi: 10.3233/BMR-2011-0277. PMID 21558611
- [Background] Jin SQ, Ding XB, Tong Y, Ren H, Chen ZX, Wang X, Li Q. Effect of saphenous nerve block for postoperative pain on knee surgery: a meta-analysis. Int J Clin Exp Med. 2015 Jan 15;8(1):368-76. eCollection 2015. PMID 25785007
- Available data/document: Study Protocol — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf#
- Available data/document: Informed Consent Form — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf#